CLINICAL TRIAL: NCT03809247
Title: Microbial Diversity of Pancreatic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, WeiWang, Chief physician, Ruijin Hospital
Other Study IDs: pancreatic diseases
Record Dates: First submitted 2018-12-24; First posted 2019-01-18 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer; Pancreatic Disease
Keywords: Pancreatic cancer; Pancreatic Disease
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Collect stool，other digestive secretions，blood and tissue samples ( (including paraffin section) and extract DNA .
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pancreatic cancer: such as Pancreatic ductal adenocarcinoma, Pancreatic acinar adenocarcinoma, and so on.
- Other pancreatic diseases: such as chronic pancreatitis, Intraductal papillary mucinous neoplasm (IPMN); Solid pseudopapillary tumors (SPT); Serous cystic neoplasm (SCN); Pancreatic neuroendocrine neoplasm (P-NN); Mucinous cystic neoplasm (MCN) and so on.

INTERVENTIONS:
Other:  — have no any intervention
  Other Names: have no any intervention

SUMMARY:
This study plans to analyze the digestive flora structure of the group of patients with pancreatic cancer.

The investigators compared the microflora of pancreatic cancer with other pancreatic diseases and healthy people，in order to obtatin the information of microbial community difference among the different groups. Finally，the investigators hope to identify the potential biomarker and pathogenic mechanisms that causes the onset and progression of pancreatic diseases.

DETAILED DESCRIPTION:
First, all the participants provided written informed consent for participating in the study. And the collecting procedures have no intervention or impact on treatment measures.

Second,the samples are collected, including the stools, the peripheral blood, and other digestive secretions. If the participants had surgical indications and received surgical treatment, the surgical resections of tissues (including paraffin section) are also collected.

Third, the participants were basically divided into three groups，cases with pancreatic cancer, cases with other pancreatic diseases, and health volunteers.

Finally, the investigators compare the microflora , its metabolites or effects among the different groups in their stool, digestive secretions, peripheral blood, pancreatic tissues ( (including paraffin section)) and so on, and hope to identify the potential biomarker and pathogenic mechanisms that causes the onset and progression of pancreatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 3 years old, ≤ 85 years old;
* After MDT discussion, routine surgery or ERCP can be performed, and the postoperative pathology is clear as pancreatic cancer and other pancreatic diseases;
* There is no serious damage to heart, liver and kidney function;

Exclusion Criteria:

* Women who are breast-feeding during pregnancy and after pregnancy;
* Patients with evidence of sensory or motor neuropathy;
* Those who have a clear cardiovascular disease, severe associated disease or active infection, including known HIV infection;
* Those who have a history of other cancers;
* Those who are allergic to drugs or their excipients

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Male / Female Age ≥ 3 years old, ≤ 85 years old;
  * After MDT discussion, routine surgery can be performed, and the postoperative pathology is clear as pancreatic cancerand other pancreatic diseases;
  * No history of antibiotics for three months before surgery, no history of yogurt containing probiotics.
  * There is no serious damage to heart, liver and kidney function.
  * After obtaining the consent and specimen collection, detailed screening found that some cases with history of antibiotics or yogurt history in three months. This part of the specimen was not discarded. As a second candidate research objects to study the effect of antibiotics or yoghurt on the flora in the disease state.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
16sRNA and metagenomics | 12/2022
  Obtain intestinal microbial information from patients with pancreatic cancer and other pancreatic diseases, and obtain information on microbial community structure, evolutionary relationships, and microbial and environmental correlations in intestinal environment samples(weight in grams).
  Correlate the patient's microbial profile with the pathogenesis of the patient to obtain biomarkers related to the pathogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Wei WANG, Dr., Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided